CLINICAL TRIAL: NCT04450758
Title: Acute Colon Resection Versus Bridge to Colon Surgery With Stent or Stoma: a Prospective Cohort Study
Brief Title: Acute Colon Resection Versus Bridge to Colon Surgery With Stent or Stoma
Acronym: ACBC
Status: Recruiting | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Pamela Buchwald, consultant colorectal surgeon, associate professor, Skane University Hospital
Other Study IDs: Skane University Hospital
Record Dates: First submitted 2020-06-14; First posted 2020-06-30 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- resection: Patients who present with obstruction due to colon cancer with a need for urgent intervention who are treated with acute resection.
- bridge to sugery: Patients who present with obstruction due to colon cancer with a need for urgent intervention who are treated with bridge to surgery i.e. either stent or stoma and resection later on.
  Interventions: Procedure: Bridge to Surgery (stent or stoma)

INTERVENTIONS:
Procedure: Bridge to Surgery (stent or stoma) — The study is an observational study and patients will not be randomized. Resection is defined as upfront surgical resection, Bridge to Surgery as a two stage procedure.
  Groups: bridge to sugery

SUMMARY:
P) patients with acute obstructive colon cancer I) resection or bridge to surgery with stent or stoma C) emergency procedure O ) morbidity and mortality within 30 days, 90 day mortality and 3 & 5 years overall survival

DETAILED DESCRIPTION:
The aim of this prospective observational study is to evaluate primary resection for malignant obstruction of the colon compared to only decompression as first intervention regarding postoperative outcomes. We hypothesize that patients with malignant obstruction benefit from avoidance of emergency cancer resection, by a two-stage procedure, with decompression by a stoma or stent as first intervention, leading to decreased short-term morbidity and mortality and improved long-term oncological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Symptomatic large bowel obstruction requiring acute intervention
* CT-verified colon obstruction due to colon cancer independent of presence of metastases
* Informed consent

Exclusion Criteria:

* Colonic perforation or bleeding
* Colonic obstruction of other origin than colon cancer
* Palliative situation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with 30-day severe morbidity | 30 days
  Clavien-Dindo >3 within 30 days postop
Overall survival after 3 years | 3 years
  survival unspecified
Number of patients with 30 day mortality | 30 days
  death within 30 days
Overall survival after 5 years | 5 years
  survival unspecified
Number of patients with 90 day mortality | 90 days
  death within 90 days

SECONDARY OUTCOMES:
Number of patients with locally radical resections | 90 days
  resections regarded as R0
Number of examined mesenteric lymph nodes | 90 days
  lymph nodes examined by pathologist
Proportion of patients receiving neoadjuvant or adjuvant treatment | 1 year
  patients receiveing chemotherapy
Proportion of patients with stomas after 3 years | 3 years
  patients with bowel continuity without stome
Recurrence rate after 3 after years | 3 years
  relapse within 3 years
Disease-free survival after 3 years | 3 years
  survival without disease relapse after 3 years
Proportion of patients not being subjected to resection of initially decompressed | 90 days
  patients not proceeding to resection
bridging interval | 90 days
  interval between stenting or stoma and resection
Number of stent complications (perforations, migration, bleeding, success rate etc) | 90 days
  complications in stent group
Number of stoma complications | 90 days
  complications in stoma group
Morbidity and survival and impact of tumour location | 5 years
  30 day morbidity and mortality depending on tumour location i.e. right or left colon
Number of laparoscopic resections | 90 days
  numbers of laparoscopic vs open resections
Number of primary anastomosis | 90 days
  number of primary anastomosis in the Bridge to Surgery vs up front resection group
Number of stomas after resection and type of stoma | 90 days
  number of stomas in Bridge to Surgery vs up front resection group
total hospital stay in days | 90 days
  days in hospital in Bridge to Surgery vs up front resection
colorectal surgeon performing resectional surgery | 90 days
  qualified colorectal surgeon, general surgeon or resident performing resectional surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Buchwald, PhD MD, Principal Investigator — Skåne University Hospital, Lund University; Tobias Axmarker, MD, Study Chair — Skåne University Hospital, Lund University
Locations (1):
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04450758/Prot_SAP_000.pdf